CLINICAL TRIAL: NCT03644459
Title: Phase I Study of the Safety, Tolerability,Pharmacokinetics and Pharmacodynamics of the Fully Humanized Anti - VEGF Monoclonal Antibody LYN00101 With Blocking of Autocrine Loops VEGFR1/2/3
Brief Title: Safety and Efficacy of the Fully Humanized Anti - VEGF Monoclonal Antibody LYN00101
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to recruit individuals for the study
Sponsor: Lynkcell Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY233-234V
Record Dates: First submitted 2018-08-03; First posted 2018-08-23 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Ovarian Cancer; Cervical Cancer; Colorectal Cancer; Stomach Cancer
Keywords: Tolerability; Safety; Humanized Anti-VEGF Monoclonal Antibody; autocrine loops; LYN00101
MeSH Terms: conditions — Ovarian Neoplasms; Uterine Cervical Neoplasms; Colorectal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LYN00101 (Experimental): Intravenous Infusion at the rate of 8 mg/kg of the patient's weight every 14 days.
  Interventions: Biological: LYN00101

INTERVENTIONS:
Biological: LYN00101 — Concentrate for intravenous infusions (10 mg / ml) with Molecular Weight 150 - 151 kDa.
  Each cycle of treatment consists of 24 weeks. Patients who enroll into this study will receive an infusion of assigned dose of LYN00101 biweekly. No intra-patient dose escalation is allowed. The proposed dose escalation sequence is 10mg/kg, starting from 8 mg/kg.

SUMMARY:
The purpose of this study is evaluate the pharmacokinetics, pharmacodynamics, immunogenicity and anti-tumor effect of of fully human anti - VEGF monoclonal antibody LY00101 and explore the potential prognostic and predictive biomarkers.

This study will not take into account the results of molecular-genetic tests of patients enrolled in the study

DETAILED DESCRIPTION:
Tumors can be inactive for years, until transformation of cells into an angiogenic phenotype occurs. This phenomenon is known as angiogenic switch. It is based on balance between inhibitors and activators of angiogenesis.

Multiple genetic changes and processes leading to malignancies, such as activation of oncogenes, can trigger angiogenic switch.

Simple diffusion of nutrients and oxygen normally occurs within not more than 1-2 mm of tumor tissue. For further growth, blood supply and development of the vasculature are necessary.

Angiogenesis level in a tumor and it's metastasis activity has correlation with density of microvessels in a primary tumor and significantly affects disease prognosis.

Angiogenesis in a body is regulated through Vascular endothelial growth factor (VEGF) and its receptors.

There is a unique binding pattern of corresponding receptors typical for all members of the VEGF family:

* VEGF-A binds with VEGFR1 and VEGFR2
* VEGF-B and PlGF bind and activate receptor VEGFR1 only
* VEGF-C and VEGF-D communicate with receptor VEGFR3 (Flt4), triggering lymphangiogenesis, and demonstrate activity correlated with VEGFR2.

According to studies, VEGFR1 binds to the ligand with the highest affinity, binding VEGF and inhibiting VEGF-mediated signaling.

The VEGF-VEGFR2 binder induces autophosphorylation (and partial dimerization) of the catalytic domain of the PI3K / v-akt signaling pathway receptor (Phosphoinositide 3-kinase / murine thymoma viral oncogene homolog - Akt or serine / threonine protein kinase B, PKB), as well as Raf and MAP2K, which further phosphorylate MAPK (Erk).

Monoclonal antibody LYN00101 is not only a potent inhibitor of VEGF, also blocks autocrine growth factor loops by inhibiting VEGF and VEGFR 1/2/3 receptors and effectively blocking neoangiogenesis.

The purpose of this study is evaluate the pharmacokinetics, pharmacodynamics, immunogenicity and anti-tumor effect of of fully human anti - VEGF monoclonal antibody LY00101 and explore the potential prognostic and predictive biomarkers.

This study will not take into account the results of molecular-genetic tests of patients enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* patients with histopathologically-documented, measurable or non measurable {evaluable}, advanced solid tumors refractory
* a life expectancy of >3 months
* ECOG performance status score of ≤ 2 at study entry
* able to provide written informed consent.
* use of effective contraceptive measures if procreative potential exists.
* an absolute neutrophil count ≥1500/mm3
* a hemoglobin level ≥ 9gm/dL
* a platelet count ≥100,000/mm3
* a total bilirubin level ≤1.5 x the ULN
* aspartate transaminase (AST) and alanine transaminase (ALT) levels ≤2.5 x the ULN or ≤5 x the ULN if known liver metastases
* adequate renal function, as defined by a serum creatinine level ≤1.5 x the ULN.

Exclusion Criteria:

* patients with any active infection (nail bed induced fungal infections were excluded), chronic infections, and tuberculosis history.
* the females were pregnant, or lactating or showed positive urine pregnancy reaction during screening.
* patients with severe heart disease, heart failure, asthma, chronic obstructive pulmonary disease or neuropsychiatric diseases.
* uncontrolled diabetes or poor compliance with hypoglycemics;
* the presence of chronically unhealed wound or ulcers
* other chronic diseases, which, in the opinion of the investigator, could compromise safety of the patient or the integrity of study.
* newly-diagnosed or symptomatic brain metastases (patients with a history of brain metastases must have received definitive surgery or radiotherapy, be clinically stable, and not taking steroids for brain edema). Anticonvulsants are allowed.
* peritoneal carcinomatosis
* pregnancy (confirmed by serum beta human chorionic gonadotropin [ßHCG]) or breast-feeding (for female patients only).
* a known history or clinical evidence of a deep vein or arterial thrombosis, or pulmonary embolism
* less than six weeks from last infusion of any anti-VEGF monoclonal antibody therapy
* known history of human immunodeficiency virus infection (HIV).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration-time curve after single dose use | up to 14 days
  Area under the concentration-time curve from 0 to ∞ with extrapolation of the final phase of the drug distribution
Peak plasma concentration after single dose use | up to 14 days
  Peak plasma concentration (Cmax) of T1h
Area under the plasma concentration after single - dose use | up to 14 days
  Area under the plasma concentration versus time curve( AUC(0-t)) of T1Hh
Elimination rate constant after single - dose use | up to 14 days
  Elimination rate constant of T1h
Time to peak after single dose use | up to 14 days
  Time to peak(Tmax) of T1h
Half time after single dose use | up to 14 days
  Half time (t1/2) of T1h
volume of distribution after single - dose use | up to 14 days
  Apparent VD - volume of distribution of T1h
Total body clearance after single-dose use | up to 14 days
  Total body clearance (CLs)of T1h
Mean residence time after single-dose use | up to 14 days
  MRT - Mean residence time of T1h
Time to peak after Each Subsequent Introduction (multiple dose) | up to 24 weeks
  Time to peak(Tmax) of T1h
Elimination rate constant after Each Subsequent Introductions (multiple dose) | up to 24 weeks
  Elimination rate constant of T1h
Area under the plasma concentration versus time curve after Each Subsequent Introduction (multiple dose) | up to 24 weeks
  Area under the plasma concentration versus time curve( AUC(0-t)) of T1Hh
Cmax of T1h after Each Subsequent Introduction (multiple dose) | up to 24 weeks
  Peak plasma concentration (Cmax) of T1h
AUC(0-∞) of T1h after Each Subsequent Introduction (multiple dose) | up to 24 weeks
  Area under the plasma concentration versus time curve(AUC(0-∞))of T1h

SECONDARY OUTCOMES:
Average plasma concentration after Each Subsequent Introduction (multiple dose) | up to 24 weeks
  Average plasma concentration in steady state/Css_avg/ of T1h
Vss of T1h after Each Subsequent Introduction (multiple dose) | up to 24 weeks
  Apparent volume of distribution in steady state /Vss/ of T1h
CT or MRI or PET/CT Control | after 8 weeks
  Tumor Necrosis and Dynamic of the Treatment ( by CT or MRI or PET/CT)
Area under the plasma concentration after each subsequent introduction (multiple dose) | up to 24 weeks
  Area under the plasma concentration versus time curve in steady state (AUCss) of T1h
Blood C-reactive protein level after Each Subsequent Introduction (multiple dose) | up to 24 weeks
  C-reactive protein/CARP/
Blood Test / morphology after Each Subsequent Introduction (multiple dose) | every week (up to 24 weeks)
  Blood Test / morphology
TNF-α level after Each Subsequent Introduction (multiple dose) | up to 24 weeks
  Tumor Necrosis Factor -alpha (TNF-α)
PGA after Each Subsequent Introduction (multiple dose) | every week up to 24 weeks
  Physician's Global Assessment /PGA/

OTHER OUTCOMES:
CLs after Each Subsequent Introduction (multiple dose) | up to 24 weeks
  Total body clearance CLs (T1h)
Apparent VD - volume of distribution of T1h after Each Subsequent Introduction (multiple dose) | up to 24 weeks
  Apparent VD - volume of distribution of T1h
Half time (t1/2) of T1h after Each Subsequent Introduction (multiple dose) | up to 24 weeks
  Half time (t1/2) of T1h